CLINICAL TRIAL: NCT06181383
Title: Phenobarbital Versus Levetiracetam Neonatal Convulsion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nashwa Nasser Heshmat, Principal Investigator, Assiut University
Other Study IDs: Phenobarbital & levetiracetam
Record Dates: First submitted 2023-11-26; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Convulsion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
If the seizure is clinically evident and prolonged, the most common first-line agent utilized is phenobarbital.(Glass et al;2016) ,Its mechanism of action is the synaptic inhibition through an action on GABA receptors, It can not only control seizures but also reduce the metabolism of the brain .(Geneva;2011) ,Phenobarbital can control 43-80% of electrical seizures (abnormal electroencephalograms) in newborns.(Sharpe et al;2020) Levetiracetam can also be used for treatment of neonatal seizures, which is safer than phenobarbital, it's mechanism of action is modulation of synaptic neurotransmitter release through binding to the synaptic vesicle protein SV2A in the brain, with less side effects on cognitive development in the levetiracetam treated subjects.(maigre et al;2013)

DETAILED DESCRIPTION:
Neonatal seizures are a commonly encountered neurologic condition in neonates.(GlassHC; 2014) They are defined as the occurrence of sudden, paroxysmal, abnormal alteration of electrographic activity at any point from birth to the end of the neonatal period.(Abend&wusthoff;2012)

Diagnoses that require priority evaluation and urgent treatment are categorized as follows:

1. Metabolic disturbances (soul;2018) as Hypoglycemia, (Hall et al;2006) ,Hypocalcemia , (Nardone et al.;2016)
2. Hypoxic conditions,( Glass et al;2016) :Hypoxic-ischemic encephalopathy ,Perinatal asphyxia
3. Intracranial hemorrhage :(Intraventricular,Intraparenchymal,Subarachnoid ,Subdural)
4. Infection :as Bacterial meningitis (Group B Streptococcus, Escherichia coli, Listeria monocytogenes)(ku at al;2015)
5. Inborn errors of metabolism - selected enzyme deficiencies :as Urea cycle defects(Yu &pearl;2013), vitamin and cofactor deficiencies: as Pyroxidine deficiency.
6. Thromboembolic: as Arterial ischemic stroke.(Govaert et al;2009) The incidence of Neonatal seizures has been reported between 1 to 5.5 per 1000 live births in term infants, with higher incidences reported in preterm infants.(Orivoli et al ;2015)

The classification of neonatal seizure types and their significant features are as follows:

1. Focal clonic seizures(Volp;1989) :Manifests as repetitive rhythmic contractions ,It can involve the face, upper or lower extremities, neck, or trunk,It cannot be extinguished by the physical suppression of movement or limb repositioning ,May migrate to other areas of the body within the same seizure (most commonly contralaterally but can occur ipsilaterally as well),If generalized, the seizure activity is diffuse, bilateral, and synchronous
2. Focal tonic seizures :Manifests as a continuous but transient extremity posturing or asymmetric posturing of the trunk or neck ,May include horizontal eye deviation ,If generalized, may mimic decerebrate posturing (upper and lower extremity tonic extension) or decorticate posturing (upper extremity flexion and lower extremity extension)
3. Myoclonic seizures(Sharma et al;2014) :Manifests as nonrepetitive contractions ,Involves flexor muscle groups of the extremity (commonly upper extremity), trunk, diaphragm, or face ,If generalized, the seizures may appear as bilateral jerking of the flexor muscles of the upper and lower extremities.
4. Subtle (unspecified) seizure is the most common type of convulsion. It includes movements such as a tremor in the eyelids; a fixed gaze in the eyes or horizontal deviation; smacking, chewing, or other oral movements; and pedaling gestures. Autonomic findings such as tachycardia andhypotension often accompany these findings.

Treatment / Management :After ensuring the patient has a patent airway, is hemodynamically stable, and has intravenous access, therapy should be targeted to treat the underlying condition identified. This can include therapeutic hypothermia for hypoxic-ischemic encephalopathy, (Papile et al ;2014) antibiotics for sepsis/meningitis, providing dextrose if the patient is severely hypoglycemic, correction of electrolyte abnormalities, or referral to neurosurgery if the patient has evidence of an intracranial hemorrhage. If the patient is suspected of having an inborn error of metabolism, halting of feeds, correcting metabolic derangements, and empiric therapy with vitamin and cofactor replacement may be initiated(Sharma&Prasad;2017) If the seizure is clinically evident and prolonged, the most common first-line agent utilized is phenobarbital.(Glass et al;2016) ,Its mechanism of action is the synaptic inhibition through an action on GABA receptors, It can not only control seizures but also reduce the metabolism of the brain .(Geneva;2011) ,Phenobarbital can control 43-80% of electrical seizures (abnormal electroencephalograms) in newborns.(Sharpe et al;2020) Levetiracetam can also be used for treatment of neonatal seizures, which is safer than phenobarbital, it's mechanism of action is modulation of synaptic neurotransmitter release through binding to the synaptic vesicle protein SV2A in the brain, with less side effects on cognitive development in the levetiracetam treated subjects.(Maitre et al;2013)

ELIGIBILITY:
Inclusion Criteria:

* All neonates with convulsions.

Exclusion Criteria:

* 1.Convulsions that occur beyond neonatal period. 2.Secondary neonatal convulsions eg: hypoglycemic, hypocalcemic, hypomagnesemic convalsions.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: Neonates present with Convulsions
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of attacks | baseline
  Phenobarbital versus levetracetam (Efficacy and safety ) in treatment of neonatal convulsion
Incidence of Possible side effects of both drugs include | baseline
  Possible side effects of both drugs include:
  * Hypotension
  * Bradycardia
  * Respiratory abnormalities
  * Sedation
  * Irritability
  * Poor feeding
  * Need of oxygen, mechanical ventilation or vasopressor medication
  * Apnea
  * Hypersensitivity reaction (angioedema, skin rash)
  * Bleeding (per gum, nose, urine)